CLINICAL TRIAL: NCT03887325
Title: To Investigate the Headache Induction and the Cerebral Hemodynamic Changes After Infusion of Maxipost in Healthy Volunteers and Migraine Patients
Brief Title: The Effects of Maxipost (BMS 204352) on Cerebral Hemodynamic and Headache in Healthy Volunteers and Migraine Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Danish Headache Center (Other)
Responsible Party: Principal Investigator, Mohammad Al-Mahdi Al-Karagholi, MD, PhD student, Principal investigator, Danish Headache Center
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Other
Other Study IDs: Maxipost P H-18052101
Record Dates: First submitted 2019-03-18; First posted 2019-03-22 (Actual); Last update posted 2020-06-16 (Actual); Status verified 2020-06

CONDITIONS: Headache, Migraine
MeSH Terms: conditions — Migraine Disorders | interventions — BMS204352; Sodium Chloride

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Maxipost (Active Comparator)
  Interventions: Drug: Maxipost
- Saline (Placebo Comparator)
  Interventions: Drug: Saline

INTERVENTIONS:
Drug: Maxipost — To investigate the role of maxipost on cerebral hemodynamic and headache in healthy volunteers and migraine patients
  Arms: Maxipost
Drug: Saline — To investigate the role of saline on cerebral hemodynamic and headache in healthy volunteers and migraine patients
  Arms: Saline

SUMMARY:
It is not previously investigated whether, there is a correlation between potassium channels and migraine, so it is unclear whether, this signaling pathway through potassium channels has an impact on migraine pathophysiology.

Maxipost (BMS 204352) is a vasoactive molecule that causes vasodilation via the big calcium dependent potassium (BKCa) channel signaling pathway. Maxipost decreases the blood pressure and maxipost infusion causes headache in healthy volunteers. A possible coherence between maxipost and headache/migraine in healthy volunteers and migraine patients is yet to be investigated.

The present study aims to clarify a possible coherence between maxipost and headache/migraine and it will help to shed light on the importance of potassium channels in migraine. In general, the study will contribute to a greater understanding of migraine pathogenesis and possibly lead to development of specific migraine treatment.

ELIGIBILITY:
Inclusion Criteria:

* Migraine patients without aura who fulfill criteria in the international classification of headaches. This does not apply to healthy volunteers.
* 18-60 years.
* 50-90 kg.
* Women of childbearing potential must use adequate contraception.

Exclusion Criteria:

* Headache less than 48 hours before the tests start
* All primary headaches, except migraine without aura for migraine patients, according to international classification of headache
* Daily consumption of drugs of any kind other than oral contraceptives
* Pregnant or nursing women.
* Cardiovascular disease of any kind, including cerebrovascular diseases.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 43 (Actual)
Dates: Start 2019-04-01 (Actual); Primary Completion 2020-02-29 (Actual); Study Completion 2020-02-29 (Actual)

PRIMARY OUTCOMES:
Occurrence and change of migraine attack | Before (-10 minutes) and after infusion (+12 hours) of maxipost compared with before and after infusion of saline
  Occurrence and of migraine according to international criteria

SECONDARY OUTCOMES:
Change in cerebral hemodynamic | Before (-10 minutes) and after infusion (+2 hours) of maxipost compared with before and after infusion of saline
  Change on velocity of media cerebri artery.
Occurrence and change of headache | Before (-10 minutes) and after infusion (+12 hours) of maxipost compared with before and after infusion of saline
  Occurrence of headache measured by numerical rating scale (NRS)
Change of diameter of the artery | Before (-10 minutes) and after infusion (+2 hours) of maxipost compared with before and after infusion of saline
  Change of diameter of superficial temporal artery and radial artery. The diameter will be measured by millimeter (mm).

CONTACTS AND LOCATIONS:
Overall Officials: Messoud A Ashina, Principal Investigator — Danish Headache Center
Locations (1):
- Danish headache center, Glostrup Municipality, Copenhagen, Denmark

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Al-Karagholi MA, Ghanizada H, Waldorff Nielsen CA, Skandarioon C, Snellman J, Lopez-Lopez C, Hansen JM, Ashina M. Opening of BKCa channels causes migraine attacks: a new downstream target for the treatment of migraine. Pain. 2021 Oct 1;162(10):2512-2520. doi: 10.1097/j.pain.0000000000002238. PMID 34252916
- [Derived] Al-Karagholi MA, Ghanizada H, Nielsen CAW, Skandarioon C, Snellman J, Lopez Lopez C, Hansen JM, Ashina M. Opening of BKCa channels alters cerebral hemodynamic and causes headache in healthy volunteers. Cephalalgia. 2020 Oct;40(11):1145-1154. doi: 10.1177/0333102420940681. Epub 2020 Aug 26. PMID 32847403